CLINICAL TRIAL: NCT03604094
Title: The Evaluation of Anatomical Variations and Dimensions of RIJV With Ultrasound in Pediatric Patients Between 0-2 Years
Brief Title: Ultrasound Measurement of RIJV in Patients Between 0-2 Years
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Filiz Uzumcugil, MD, Asist. Prof., Hacettepe University
Other Study IDs: Ultrasonography of RIJV
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Anatomic Abnormality; Internal Jugular Vein; Neonates; Infants, Premature; Children
Keywords: central venous catheter, pediatrics, ultrasound imaging
MeSH Terms: conditions — Congenital Abnormalities; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: 0-1 month old newborns
  Interventions: Procedure: Ultrasonographic evaluation
- Group II: 1 month-2 year-old pediatric patients
  Interventions: Procedure: Ultrasonographic evaluation

INTERVENTIONS:
Procedure: Ultrasonographic evaluation — Right internal jugular vein will be evaluated with ultrasound for anatomical variations and dimensions

SUMMARY:
After obtaining parental consent ultrasonographic evaluation of right internal jugular vein will be performed in pediatric patients undergoing elective surgeries between 0-2 years of age. The patients for whom central venous catheterization is indicated will be included. The success rates and outcomes of catheterization will be recorded.

ELIGIBILITY:
Inclusion Criteria:

0-2 years Elective surgery Requirement for central venous cannulation

Exclusion Criteria:

Congenital cardiovascular anomalies Emergency surgeries Previous cannulation or any intervention on the neck

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy 0-2 year-old patients undergoing elective surgery.
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Anatomical variations and dimensions of right internal jugular vein | 1 year
  The central vein will be evaluated by ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Filiz Uzumcugil, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No